CLINICAL TRIAL: NCT04802499
Title: Investigation of the Validity and Reliability of the Turkish Version of Telehealth Satisfaction Survey (TeSS)
Brief Title: Turkish Version of Telehealth Satisfaction Survey (TeSS)
Status: Completed | Type: Observational
Sponsor: Mustafa Kemal University (Other)
Responsible Party: Principal Investigator, Irem Hüzmeli, Phd lecturer, Mustafa Kemal University
Other Study IDs: HatayMKU
Record Dates: First submitted 2021-03-14; First posted 2021-03-17 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: Healthy; Health, Subjective; Health Knowledge, Attitudes, Practice
Keywords: telehealth; satisfication; telerehabilitation
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 15 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- persons who using telehealth (patients): patients who have received telehealth
  Interventions: Procedure: Turkish Reliability and Validity of TESS
- caregivers: family member of the patients who recieved telehealth
  Interventions: Procedure: Turkish Reliability and Validity of TESS
- health professions: persons who use the telehealth.
  Interventions: Procedure: Turkish Reliability and Validity of TESS

INTERVENTIONS:
Procedure: Turkish Reliability and Validity of TESS — Translation and cultural adaptation of the scale will be designed according to the appropriate procedure. Turkish data will be uploaded in the online online method. The scale will be communicated online to those who have received telerehabilitation services, caregivers and healthcare professionals who have applied it. The reliability of the questionnaire will be made by test-retest and internal consistency analysis. Volunteers will be asked to answer the questionnaire online after 5 days. After two weeks, the participants will be asked to answer the questionnaire again with the same method online with 5 days intervals. After all data are collected, validity analysis will be performed

SUMMARY:
The Turkish validity and reliability of the scale, which was created to evaluate the satisfaction of individuals, caregivers, and coordinator providing telerehabilitation services within the scope of telehealth, will be investigated.

DETAILED DESCRIPTION:
The telehealth satisfaction survey (TeSS) has been developed according to expectations, taking into account a device previously used in telehealth studies in Saskatchewan. The scale was initially used as part of a national study to evaluate the use of telehealth practices in improving professional access by residents of isolated Northern First Nations communities.The scale designed for telehealth services has been developed in English. Validity and reliability studies have been carried out by being translated into various languages. The Turkish validity and reliability study of the scale, originally in English, has not been conducted before.

ELIGIBILITY:
Inclusion Criteria:

* Men and woman who used telehealth

Exclusion Criteria:

* Individuals who have the poor cooperation Mini-Mental State Exam scores of under 23

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: telehealth patients caregivers and health professionals who practice telehealth
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2021-03-12 (Actual); Primary Completion 2022-05-12 (Actual); Study Completion 2022-06-12 (Actual)

PRIMARY OUTCOMES:
Turkish Reliability and Validity of TESS (telehealth Satisfaction Survey) for patients, caregivers and health professional who use telehealth | March 2021-April 2022
  validation and reliability of survey in Turkish

CONTACTS AND LOCATIONS:
Overall Officials: Irem Huzmeli, PhD, Study Director — Mustafa Kemal University
Locations (1):
- Hatay Mustafa Kemal University, Hatay, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No